CLINICAL TRIAL: NCT05692206
Title: In Chronic Neck Pain; Kinesiophobia, Neck Awareness Examination of Cognitive and Cognitive Functions at Different Levels of Functionality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Yunus Ozkaya, Physiotherapist, Mustafa Kemal University
Other Study IDs: MustafaKUYO
Record Dates: First submitted 2022-12-21; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- according to the neck disability index, mildly and moderately affected
  Interventions: Other: evaluation
- According to the neck disability index, severely affected and very severely affected
  Interventions: Other: evaluation

INTERVENTIONS:
Other: evaluation — Surveys will be administered to the participants. Participants will be given a stroop TBAG test.

SUMMARY:
Chronic neck pain is a common problem in our society. With the Neck Disability Index, we can classify the functional status of individuals with chronic neck pain as "no restriction, mildly limited, moderately limited, severely restricted, completely limited". In this study, the difference between cognitive functions, kinesiophobia and neck awareness between those who have a functional status according to the Neck Disability Index and those whose functional status is "slightly limited-moderately restricted" and those who are "severely limited-totally limited" will be investigated with questionnaires and evaluations. The study will provide information about whether there is a difference between individuals with chronic neck pain regarding cognitive functions, kinesiophobia and neck awareness according to their functional status. Thus, it will contribute to the literature to provide clinicians with awareness about the functionality levels in chronic neck pain and to consider individuals within this framework.

DETAILED DESCRIPTION:
Neck pain is a health problem that individuals experience at least once in their lives and that happens to approximately 43% of individuals. Neck pain is the most common chronic pain after chronic low back pain. Situations such as physical strains during any activity, staying in a static posture for a long time, using an inappropriate bag or carrying a weight that forces the individual can affect the structures such as joints, discs, ligaments, and muscles in the cervical region and cause pain. It should not be forgotten that the symptoms seen in individuals with neck pain can be seen to go away on their own within a few weeks, and up to 30% of them can become chronic. Considering that neck pain can become chronic, it will be understood that the physiological and psychological effects of this chronic neck pain on individuals must be evaluated. For this reason, it would be appropriate to evaluate not only the pain but also the functional status in accordance with the biopsychosocial model with special approaches for individuals suffering from chronic neck pain.

Chronic neck pain negatively affects the daily living activities of individuals and causes disability as well as functional limitations. The fact that deaths from neck pain are very rare in general ensures that the main goal of treatment is to improve functional status. For an appropriate and effective treatment planning for individuals, it is necessary to analyze the current functional status of the individual well and to understand which factors affect their functional status.

Recent studies have shown that pain and disability are directly proportional to the increase in degeneration in individuals with chronic neck pain. It was concluded that this ratio was accompanied by physical activities and general health status.

Long sitting times, working conditions, unconscious use of technology, which we often encounter in our daily lives, cause individuals to be physically inactive and lead a sedentary life. In addition, postural problems, decrease in muscle quantity and strength, obesity, chronic diseases, and diseases such as cancer can negatively affect our health in our future lives. These conditions negatively affect the physical health of the society and may also lead to regression in cognitive functions. Psychological variables were also associated with neck pain from the initial stage of neck pain to its chronic stages. Cognitive factors, depression, anxiety and related emotional states are associated with pain and disability and are determinant risk factors for chronic neck pain and disability. Sebastian et al. emphasize that it is important to evaluate certain cognitive abilities at all ages, not just in childhood or old age, in order to observe changes that occur throughout life.

In a study examining the relationship between pain, quality of life and kinesiophobia in nonspecific chronic neck pain, it was determined that patients with chronic neck pain had kinesiophobia. At the end of a study by Demirbüken et al., it was seen that 80.2% of the individuals participating in the study had a high level of fear of movement.

In a disorder in the neck region, muscle dysfunction occurs as a result of pain, disruption of sensory-motor input, and the transfer of the function of the deep muscles to the superficial muscles. These problems can cause the neck to be perceived as asymmetrical, tense, oversized or small, and its position and movement abnormal. In order to eliminate problems such as pain, tension, asymmetry, and deterioration of position-motion perception, it is important for physiotherapists to evaluate and treat in-body and extra-body awareness, and to raise body awareness to a conscious level.

As a result, the results obtained by examining cognitive functions, kinesiophobia and neck awareness according to the affect status of individuals with chronic neck pain are important for individuals to overcome this process quickly and healthily. This study is interesting with its support for an effective treatment and its contribution to the literature.

The study will be carried out with individuals who apply to Malatya Kanalboyu Physical Therapy and Rehabilitation Center with the complaint of chronic neck pain, who meet the inclusion criteria. By examining previous studies, this study was planned to be carried out on 100 people. Demographic information (name, surname, age, gender, telephone) of the individuals participating in the study will be taken.

Neck Disability Index questionnaire will be applied to determine the functionality levels of individuals. The Neck Disability Questionnaire consists of 10 questions related to pain intensity, personal care, lifting, reading, concentration, headache, working, driving, sleeping and recreational activities. There are 6 options for each question, ranging from 0 to 5 points. 0 points means no restrictions, 50 points means full apology. A score of 0-4 means no restriction, a score of 5-14 means mildly restricted, a score of 15-24 moderately restricted, 25-34 severely restricted, and 35 and above means completely restricted. In our study, those with mild and moderate restraints will form the 1st group, and those with severe and complete restraint will form the 2nd group.

Stroop TBAG test will be applied to evaluate cognitive functions. Stroop TBAG Test; It is designed to measure the perceptual setup, the ability to adjust itself to the desired demand under the influence of distraction, the ability to rule out a habitual behavioral movement, and the focusing skills of individuals. The test consists of 5 separate parts in total. From the patient; On the first paper, the words written in black are asked to be read. He is asked to read the words written in color on the second piece of paper. On the third piece of paper, it is asked to say the colors of the circle shapes. On the fourth paper, only the color is asked to be said without reading the unrelated words written in color. On the fifth piece of paper, he is asked to correctly say the color of the words printed in a different color than his own.

Standardized Minimental Test will be applied for cognitive function evaluation. This test consists of five parts: orientation, recording, attention and calculation, recall and language tests. The total score is 30, those who score 24 points or less are at risk for cognitive impairment. A total score of 17 or less is considered severe, a score between 18-23 is considered a moderate disorder, and a score of 24 and above is considered normal.

Tampa Kinesiophobia Scale will be used to measure fear of movement (kinesiophobia). The purpose of developing this scale is to distinguish patients with normal response and high fear of movement. There are 17 questions in the scale and a 4-point Likert scoring is used. After the 4, 8, 12 and 16 items are reversed in the scoring, a total score is calculated and a minimum of 17 and a maximum of 68 points are obtained. The higher the score on the scale, the greater the fear of movement.

The Fremantle Neck Awareness Questionnaire will be used to measure the neck awareness of the individuals participating in the study. The questionnaire asks individuals 9 questions such as how they perceive their neck relative to their body, how they perceive their body position. Likert type assessing individual-specific altered perception (0 = Never/Never feel this way, 1 = I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I feel this way often, 4 = I feel this way all or most of the time) It's a simple survey.

ELIGIBILITY:
Inclusion Criteria:

* A score of 24 or higher on the Standardized Minimental Test.
* Having chronic neck pain problem for the last 6 months.
* Being between the ages of 40-59.
* Volunteer to participate in the study.
* To be able to read and write.

Exclusion Criteria:

* To have a score of 0-4 from the Neck Disability Questionnaire.
* Having undergone musculoskeletal surgery.
* Having a rheumatic or neurological disease.
* pregnancy status
* Having a congenital musculoskeletal disorder.
* The presence of trauma, infectious pathology or scoliosis affecting the spine.
* Any visual impairment.

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: According to the neck disability index, those with mild and moderate severity will be determined as the first group, and those who are severely and severely affected will be determined as the second group.
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2023-02-13 (Estimated); Primary Completion 2023-04-07 (Estimated); Study Completion 2023-04-07 (Estimated)

PRIMARY OUTCOMES:
cognitive functions | 8 week
  Stroop TBAG test will be applied to evaluate cognitive functions. Stroop TBAG Test; It is designed to measure the perceptual setup, the ability to adjust itself to the desired demand under the influence of distraction, the ability to rule out a habitual behavioral movement, and the focusing skills of individuals. The test consists of 5 separate parts in total. The patient reads the words written in black on the first sheet of paper. The patient reads the words written in color on the second sheet of paper. The patient tells the colors of the circle shapes on the third sheet of paper. The patient simply says the color of the fourth sheet without reading the unrelated words written in color. The patient correctly tells the color of the words printed in a different color from his own color on the fifth paper.
kinesiophobia | 8 week
  Tampa Kinesiophobia Scale will be used to measure fear of movement (kinesiophobia). The purpose of developing this scale is to distinguish patients with normal response and high fear of movement. There are 17 questions in the scale and a 4-point Likert scoring is used. After the 4th, 8th, 12th and 16th items are reversed in scoring, a total score is calculated and a minimum of 17 and a maximum of 68 points are obtained. The higher the score on the scale, the greater the fear of movement.
neck awareness | 8 week
  The Fremantle Neck Awareness Questionnaire will be used to measure the neck awareness of the individuals participating in the study. The questionnaire asks individuals 9 questions such as how they perceive their neck relative to their body, how they perceive their body position. Likert type assessing individual-specific altered perception (0 = Never/Never feel this way, 1 = I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I feel this way often, 4 = I feel this way all or most of the time) it is a simple survey.
Neck Disability Index | 8 week
  The Neck Disability Questionnaire consists of 10 questions related to pain intensity, personal care, lifting, reading, concentration, headache, working, driving, sleeping and recreational activities. There are 6 options for each question, ranging from 0 to 5 points. 0 points means no restrictions, 50 points means full apology. A score of 0-4 means no restriction, a score of 5-14 means mildly restricted, a score of 15-24 moderately restricted, 25-34 severely restricted, and 35 and above means completely restricted.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunus Özkaya, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No